CLINICAL TRIAL: NCT05018832
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for the Treatment of Traumatic Brain Injury
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for TBI
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-20-ATG-12-4
Record Dates: First submitted 2021-08-20; First posted 2021-08-24 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; stem cell treatment
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (AlloRx) (Experimental): Single intravenous infusion of 100 million cells
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells for the treatment of traumatic brain injury

DETAILED DESCRIPTION:
Studies have shown that stem cell treatment is safe and efficacious for the treatment of Traumatic brain injury (TBI). This patient funded trial aims to study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells (UC-MSCs) for the treatment of TBI. Patients with TBI will receive a single intravenous infusion of UC-MSCs. The total dose will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of traumatic brain injury
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur
* Seizure disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (1):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang S, Cheng H, Dai G, Wang X, Hua R, Liu X, Wang P, Chen G, Yue W, An Y. Umbilical cord mesenchymal stem cell transplantation significantly improves neurological function in patients with sequelae of traumatic brain injury. Brain Res. 2013 Sep 26;1532:76-84. doi: 10.1016/j.brainres.2013.08.001. Epub 2013 Aug 11. PMID 23942181
- [Background] Tian C, Wang X, Wang X, Wang L, Wang X, Wu S, Wan Z. Autologous bone marrow mesenchymal stem cell therapy in the subacute stage of traumatic brain injury by lumbar puncture. Exp Clin Transplant. 2013 Apr;11(2):176-81. doi: 10.6002/ect.2012.0053. Epub 2012 Aug 11. PMID 22891928
- [Background] Wang Z, Luo Y, Chen L, Liang W. Safety of neural stem cell transplantation in patients with severe traumatic brain injury. Exp Ther Med. 2017 Jun;13(6):3613-3618. doi: 10.3892/etm.2017.4423. Epub 2017 May 4. PMID 28588689